CLINICAL TRIAL: NCT07301138
Title: A Prospective Study of BEBT-908 in Combination With Chemotherapy for Patients With MEF2D-Rearranged and Pre-B Acute Lymphoblastic Leukemia in Complete Remission With Minimal Residual Disease Positivity
Brief Title: BEBT-908 Plus Chemotherapy Treatment for CR MRD-Positive MEF2D-Rearranged and Pre-B Acute Lymphoblastic Leukemia Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, chief physician, MD, PhD, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-ALL 2025-B04
Record Dates: First submitted 2025-12-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Pre-B acute lymphoblastic leukemia; MEF2D-rearranged; Minimal Residual Disease; BEBT-908
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — BEBT-908; Cyclophosphamide; Vincristine; Dexamethasone; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): * BEBT-908 for Injection, dosage of administration:12.3mg/m2，frequency and duration of administration: on the 1st,3rd,5th,8th, 10th and 12th days of each cycle and 28 days as a cycle.
  * Cyclophosphamide Injection, dosage of administration: 150 mg/m2 every 12 hours on days 1 to 3 of odd cycles, and 28 days as a cycle.
  * Vincristine Injection, dosage of administration: 1.4mg/m2 on day 4 and 11 of odd cycles, and 28 days as a cycle.
  * Dexamethasone Injection, dosage of administration: 20 mg per day on days 1 to 4 and 11 to 14 of odd cycles, and 28 days as a cycle.
  * Methotrexate Injection, dosage of administration: 1g/m2 on day 1 of even cycles, and 28 days as a cycle.
  * Cytarabine Injection, dosage of administration: 0.5 g/m2 given every 12 hours on day 2 and 3 of even cycles, and 28 days as a cycle.
  Interventions: Drug: BEBT-908; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Dexamethasone; Drug: Methotrexate; Drug: Cytarabine

INTERVENTIONS:
Drug: BEBT-908 — BEBT-908 for Injection, dosage of administration: 12.3mg/m2，frequency and duration of administration: on the 1st,3rd,5th,8th,10th and 12th days of each cycle, and 28 days as a cycle.
Drug: Cyclophosphamide — Cyclophosphamide Injection, dosage of administration: 150 mg/m2 every 12 hours on days 1 to 3 of odd cycles, and 28 days as a cycle.
Drug: Vincristine — Vincristine Injection, dosage of administration: 1.4mg/m2 on day 4 and 11 of odd cycles, and 28 days as a cycle.
Drug: Dexamethasone — Dexamethasone Injection, dosage of administration: 20 mg per day on days 1 to 4 and 11 to 14 of odd cycles, and 28 days as a cycle.
Drug: Methotrexate — Methotrexate Injection, dosage of administration: 1g/m2 on day 1 of even cycles, and 28 days as a cycle.
Drug: Cytarabine — Cytarabine Injection, dosage of administration: 0.5 g/m2 given every 12 hours on day 2 and 3 of even cycles, and 28 days as a cycle.

SUMMARY:
This investigator-initiated, prospective, single-arm, multicenter clinical trial aims to evaluate the efficacy and safety of BEBT-908 (a HDAC/PI3Kα inhibitor provided by BeBetter Med Inc ,Guangzhou, China) combined with chemotherapy in patients with MEF2D-rearranged and pre-B acute lymphoblastic leukemia who are in complete remission (CR) but remain minimal residual disease (MRD) positive.

DETAILED DESCRIPTION:
MEF2D-rearranged and pre-B acute lymphoblastic leukemia patients achieving CR after chemotherapy and have MRD+ will be given BEBT-908 (12.3 mg/m2) combined with Mini-Hyper-CVD and Mini-MTX/Ara-C chemotherapy for two cycles.

After two cycles, If MRD negativity is achieved and the patient is eligible for transplantation, hematopoietic stem cell transplantation will be performed; if MRD negativity is achieved but the patient is not suitable for transplantation, an additional six courses of BEBT-908-based combination chemotherapy will be given. Patients who fail to reach MRD negativity will be withdrawn from the study.

A total of 23 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily agrees to participate in this trial and signs the informed consent form, and is able to understand and comply with all study requirements;
2. Age between ≥18 and ≤75 years at screening, with no gender restrictions;
3. Meets the diagnostic criteria for BCP-ALL (according to the 2022 WHO classification) and fulfills any one of the following conditions:

1) Positive for MEF2D rearrangement 2) Philadelphia chromosome negative and consistent with a Pre-B immunophenotype (according to the EGIL 1995 immunophenotyping criteria, cytoplasmic IgM+); 4. Diagnosed with BCP-ALL in complete remission but with positive minimal residual disease (MRD), defined as: achieving hematologic complete remission (CR) after treatment (bone marrow blast count <5% by morphology) but with positive MRD (MRD ≥10-⁴, as detected by flow cytometry and/or PCR); 5. ECOG performance status score of 0-2 at screening; 6. Expected survival is more than 3 months. 7. Satisfactory organ function, meeting the following criteria:

1. Serum creatinine ≤1.5 times the upper limit of normal（ULN）；
2. Left ventricular ejection fraction (LVEF) >50%; 3）Total bilirubin ≤2 times ULN；Alanine aminotransferase (ALT) ≤3 times ULN; Aspartate aminotransferase (AST) ≤3 times ULN

Exclusion Criteria:

1. Known allergy to the study drug or its excipients.
2. Presence of severe and/or uncontrolled infection.
3. Severe cardiac disease, including: heart failure classified as New York Heart Association (NYHA) functional class III or IV; history of acute myocardial infarction within 6 months prior to screening; uncontrolled arrhythmias or electrophysiological abnormalities such as sick sinus syndrome, third degree atrioventricular block, QTc > 480 ms, ventricular tachycardia, persistent atrial fibrillation with rapid ventricular response, etc.; or severe structural cardiac abnormalities on echocardiography or left ventricular ejection fraction (LVEF) < 50 %.
4. Primary central nervous system diseases, including cerebrovascular accident, intracranial infection, etc., within six months before screening.
5. Severe primary pulmonary diseases, including significant impairment of pulmonary ventilation/diffusion function, respiratory failure, etc.
6. Severe hepatic impairment: total bilirubin (TB), gamma glutamyl transferase (γGT), ALT, or AST > 3 times ULN at baseline or after hepatoprotective therapy; or conditions such as severe hepatitis, cirrhosis, etc.
7. Severe renal impairment: serum creatinine > 1.5 × ULN; or uncorrected acute kidney injury.
8. Acute or chronic pancreatitis, with serum amylase > 3 × ULN.
9. Pregnancy or lactation.
10. History of other prior malignancies that may affect protocol compliance or interpretation of study results.
11. Diagnosed major psychiatric disorder or predisposition to psychiatric illness that would significantly impair the ability to participate in the clinical study.
12. Any other condition deemed by the investigator as unsuitable for study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MRD negativity rate | At the end of Cycle 2 of BEBT-908 combined chemotherapy treatment (each cycle is 28 days)
  The proportion of patients who reach MRD negative

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months
  Interval from the date of the feedback to the time of death due to any reason
Relapse-free survival (RFS) | up to 24 months
  Interval from the date of BEBT-908 treatment to the time of diagnosis of hematological recurrence or death from any cause
Progression-Free Survival (PFS) | up to 24 months
  Interval from the date of BEBT-908 treatment to the time of diagnosis of disease progression or death from any cause
Incidence of adverse events | up to 24 months
  The proportion of patients who have adverse events after BEBT-908 treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China